CLINICAL TRIAL: NCT07311707
Title: A Randomized Controlled Trial Comparing Primary Closure Versus Open Surgical Technique in the Management of Pilonidal Sinus Disease
Brief Title: Primary Closure vs Open Technique for Pilonidal Sinus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Dr Asghar Ali, Principal Investigator, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 153/DME/KMC
Record Dates: First submitted 2025-12-12; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pilonidal Sinus Disease; Sacrococcygeal Pilonidal Sinus; Chronic Infected Sinus Tract; Post-surgical Wound Healing
Keywords: Pilonidal Sinus; Primary Closure; Wound Healing; Randomized Controlled Trial; Surgical Site Infection
MeSH Terms: conditions — Pilonidal Sinus; Surgical Wound Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Excision with Primary Closure (Experimental): Participants assigned to this arm will undergo complete surgical excision of the pilonidal sinus tract followed by primary closure of the wound using standard suturing techniques. All procedures will be performed by an experienced surgical team. Postoperative management will be standardized and will include routine wound care, sitz baths, and antibiotic prophylaxis according to institutional protocol. Participants will be followed postoperatively to assess wound healing progress, postoperative complications, and recurrence during scheduled follow-up visits.
  Interventions: Procedure: Primary Suturing of Surgical Wound; Procedure: Open Surgical Wound Management
- Excision with Open (Lay-Open) Technique (Experimental): Participants assigned to this arm will undergo complete surgical excision of the pilonidal sinus tract, with the wound left open to heal by secondary intention. Standard postoperative wound care will be provided, including regular dressings, sitz baths, and antibiotic prophylaxis according to institutional protocol. Participants will be monitored during follow-up visits to assess wound healing, postoperative complications, and recurrence.
  Interventions: Procedure: Primary Suturing of Surgical Wound; Procedure: Open Surgical Wound Management

INTERVENTIONS:
Procedure: Primary Suturing of Surgical Wound — The surgical site will be closed immediately after surgery using standard suturing techniques to approximate wound edges. This is the conventional method for wound closure in this study.
Procedure: Open Surgical Wound Management — The surgical site will be managed using an open approach without primary closure, with standard postoperative wound care.

SUMMARY:
The purpose of this randomized controlled trial is to compare two commonly used surgical techniques for the treatment of pilonidal sinus disease: excision with primary closure and excision with open (lay-open) technique. Pilonidal sinus disease is a chronic inflammatory condition of the natal cleft that causes pain, discharge, and functional discomfort, particularly in young adults.

The primary aim of the study is to evaluate whether excision followed by primary closure leads to faster wound healing compared to the open surgical technique. Secondary aims include comparing postoperative wound infection and recurrence rates between the two surgical approaches.

Eligible participants aged 20 to 50 years with uncomplicated pilonidal sinus disease will be randomly allocated to one of two treatment groups. All surgical procedures will be performed by an experienced surgical team at Khyber Teaching Hospital, Peshawar. Postoperative care and follow-up schedules will be standardized for all participants. Outcomes will be assessed during follow-up visits at 1 week, 3 weeks, and 12 weeks after surgery.

This study is intended to provide evidence to guide surgical decision-making and improve postoperative outcomes for patients with pilonidal sinus disease.

DETAILED DESCRIPTION:
Background and Rationale

Pilonidal sinus disease is a chronic inflammatory condition that primarily affects the natal cleft region and is most commonly seen in young adults. The disease is characterized by pain, discharge, recurrent infection, and limitations in daily activities, resulting in a reduced quality of life. It is more frequently observed in males and in individuals with prolonged sitting habits, obesity, or excessive body hair.

The pathogenesis of pilonidal sinus disease is widely accepted to be acquired, involving the penetration of loose hairs into the skin of the natal cleft, followed by a foreign body reaction and secondary infection. Surgical management remains the definitive treatment option, aiming to excise diseased tissue, promote wound healing, minimize complications, and reduce recurrence.

Multiple surgical techniques have been described in the literature; however, there is no universally accepted standard approach. Excision with primary closure allows immediate wound closure and potentially faster recovery, while excision with open (lay-open) technique permits healing by secondary intention and may reduce recurrence in certain cases. Variability in outcomes reported across studies highlights the need for randomized controlled trials conducted within uniform clinical settings.

This study is designed to compare these two surgical techniques under standardized operative and postoperative conditions in order to evaluate their relative effectiveness.

Study Objectives

Primary Objective To compare wound healing time between excision with primary closure and excision with open (lay-open) technique in patients with pilonidal sinus disease.

Secondary Objectives To compare the frequency of postoperative wound infection between the two surgical techniques.

To compare the rate of recurrence within the follow-up period between the two surgical techniques.

Study Design This study is a single-center, parallel-group, randomized controlled trial conducted at the Department of Surgery, Khyber Teaching Hospital, Peshawar, Pakistan. Participants will be randomly assigned in a 1:1 ratio to one of two intervention groups using a computer-generated block randomization method.

The study will be conducted in accordance with institutional ethical guidelines, and written informed consent will be obtained from all participants prior to enrollment.

Study Population Adult male and female patients aged 20 to 50 years diagnosed with uncomplicated pilonidal sinus disease will be assessed for eligibility.

Eligibility criteria, outcome measures, and follow-up schedules are defined in their respective sections of the record and are not duplicated here.

Sample Size and Sampling Technique A total sample size of 132 participants (66 per group) was calculated using the WHO sample size calculator, assuming a 95% confidence level, 80% power, and reference values from previously published studies. Eligible patients meeting inclusion criteria will be recruited using a non-probability consecutive sampling technique until the required sample size is achieved.

Randomization and Allocation Participants will be randomly allocated to one of the two study groups using computer-generated block randomization. Allocation concealment will be ensured through sealed opaque envelopes opened at the time of surgery.

Intervention Details All surgical procedures will be performed by the same surgical team with adequate experience to minimize inter-operator variability.

Group A: Excision with Primary Closure Complete excision of the pilonidal sinus tract will be performed, followed by primary wound closure using sutures after achieving adequate hemostasis.

Group B: Excision with Open (Lay-Open) Technique The pilonidal sinus tract and surrounding affected tissue will be excised, and the wound will be left open to heal by secondary intention with regular postoperative dressings.

All participants will receive standardized postoperative care, including wound dressing protocols, sitz baths, and antibiotic prophylaxis as per institutional guidelines.

Follow-up and Outcome Assessment

Participants will be evaluated postoperatively at:

1 week 3 weeks 12 weeks

Assessments will focus on wound healing status, signs of infection, and clinical evidence of recurrence. Data will be recorded using a standardized proforma by the principal investigator.

Statistical Analysis Data analysis will be performed using SPSS version 22. Quantitative variables will be summarized as mean and standard deviation, while qualitative variables will be presented as frequencies and percentages. Appropriate statistical tests will be applied to compare outcomes between groups, and a p-value of less than 0.05 will be considered statistically significant.

Key Words Pilonidal sinus disease, Primary closure, Open surgical technique, Wound healing, Wound infection, Recurrence, Randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 20 to 50 years.

Clinically diagnosed with pilonidal sinus (persistent painful discharging wound in the buttock cleft for more than eight weeks, VAS >4).

Patients willing to provide written informed consent.

Exclusion Criteria:

* Pilonidal sinus located away from the midline coccyx.

Presence of abscess formation.

Patients with underlying conditions affecting wound healing (e.g., diabetes mellitus).

Recurrent pilonidal sinus.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Duration of Wound Healing After Surgery | 12 weeks
  Time (in days) from surgical intervention to complete wound epithelialization, assessed at 1, 3, and 12 weeks postoperatively, comparing primary closure versus open surgical technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Wasim Khan, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: No